CLINICAL TRIAL: NCT00096720
Title: Investigating Effects of Short-term Treatment With Pramipexole or Levodopa on [123I]B-CIT and SPECT Imaging in Early Parkinson's
Brief Title: Study of the Effects of Dopaminergic Medications on Dopamine Transporter Imaging in Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: Boehringer Ingelheim (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Danna Jennings M.D., Institute for Neurodegenerative Disorders
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: INSPECT
Record Dates: First submitted 2004-11-12; First posted 2004-11-15 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2007-05

CONDITIONS: Parkinson Disease; Parkinsonian Syndrome
Keywords: parkinson; brain imaging; diagnosis
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Disease | interventions — Levodopa; Pramipexole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: levodopa
Drug: Mirapex (pramipexole)
Procedure: [123I]ß-CIT and SPECT imaging

SUMMARY:
Study participants who have been clinically diagnosed with Parkinson disease will receive no treatment, treatment with either levodopa, or treatment with Mirapex for a period of 12 weeks. Over the course of the study subjects will travel to the Institute for Neurodegenerative Disorders (IND) in New Haven, Connecticut for brain imaging.

DETAILED DESCRIPTION:
Brain imaging will be conducted three times during this study. Study participants will travel to IND for [123I]ß-CIT and SPECT imaging (scan 1). Subjects will be randomized to no treatment, treatment with either levodopa, or treatment with Mirapex and undergo treatment for a period of 12 weeks. Subjects will return to IND for [123I]ß-CIT and SPECT imaging (scan 2) after 12 weeks of treatment and withdraw from the medication following the scan. Eight to 12 weeks after medication withdrawal, a final [123I]ß-CIT and SPECT imaging study (scan 3) will be performed at IND. The imaging outcome, striatal uptake of [123I]ß-CIT, from scan 1 (untreated) and scan 2 (treated with levodopa or pramipexole) will be compared to determine if there is a significant change in the uptake of the marker that may be attributed to levodopa or pramipexole treatment. In addition, scan 3 will be compared to scan 2 to determine the duration and reversibility of any regulatory effect that occurs. The subjects will be randomized, but not blinded to study drug assignment. The imaging technologist and all imaging analyses will be performed by investigators blinded to study drug assignment.

ELIGIBILITY:
Inclusion Criteria:

* 30 years or older at time of Parkinson Disease (PD) diagnosis
* clinical diagnosis of PD of equal to or less than 7.5 years
* Normal laboratory screening

Exclusion Criteria:

* Participant is pregnant
* Participant has atypical or drug induced PD
* Participant has significant dementia

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2004-02; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change in outcomes from scan 1 to scan 2

SECONDARY OUTCOMES:
Change in outcomes from scan 2 to scan 3

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (13):
- United States (13):
  - Pacific Neuroscience Medical Group, Oxnard, California
  - Colorado Neurology, PC, Englewood, Colorado
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - University of Florida Movement Disorders Center, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - RUSH University Medical Center, Chicago, Illinois
  - Boston University Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Parkinson's Disease and Movement Disorders Center of Albany Medical College, Albany, New York
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - NeuroHealth, Inc., Warwick, Rhode Island
  - University of Tennessee Health Science Center, Memphis, Tennessee

REFERENCES:
- [Background] Ahlskog JE. Slowing Parkinson's disease progression: recent dopamine agonist trials. Neurology. 2003 Feb 11;60(3):381-9. doi: 10.1212/01.wnl.0000044047.58984.2f. PMID 12580184
- [Background] Ahlskog JE, Uitti RJ, O'Connor MK, Maraganore DM, Matsumoto JY, Stark KF, Turk MF, Burnett OL. The effect of dopamine agonist therapy on dopamine transporter imaging in Parkinson's disease. Mov Disord. 1999 Nov;14(6):940-6. doi: 10.1002/1531-8257(199911)14:63.0.co;2-y. PMID 10584667
- [Background] Brucke T, Asenbaum S, Pirker W, Djamshidian S, Wenger S, Wober C, Muller C, Podreka I. Measurement of the dopaminergic degeneration in Parkinson's disease with [123I] beta-CIT and SPECT. Correlation with clinical findings and comparison with multiple system atrophy and progressive supranuclear palsy. J Neural Transm Suppl. 1997;50:9-24. PMID 9120429
- [Background] Fahn S. Is levodopa toxic? Neurology. 1996 Dec;47(6 Suppl 3):S184-95. doi: 10.1212/wnl.47.6_suppl_3.184s. No abstract available. PMID 8959987
- [Background] Guttman M, Stewart D, Hussey D, Wilson A, Houle S, Kish S. Influence of L-dopa and pramipexole on striatal dopamine transporter in early PD. Neurology. 2001 Jun 12;56(11):1559-64. doi: 10.1212/wnl.56.11.1559. PMID 11402115
- [Background] Innis RB, Seibyl JP, Scanley BE, Laruelle M, Abi-Dargham A, Wallace E, Baldwin RM, Zea-Ponce Y, Zoghbi S, Wang S, et al. Single photon emission computed tomographic imaging demonstrates loss of striatal dopamine transporters in Parkinson disease. Proc Natl Acad Sci U S A. 1993 Dec 15;90(24):11965-9. doi: 10.1073/pnas.90.24.11965. PMID 8265656
- [Background] Innis RB, Marek KL, Sheff K, Zoghbi S, Castronuovo J, Feigin A, Seibyl JP. Effect of treatment with L-dopa/carbidopa or L-selegiline on striatal dopamine transporter SPECT imaging with [123I]beta-CIT. Mov Disord. 1999 May;14(3):436-42. doi: 10.1002/1531-8257(199905)14:33.0.co;2-j. PMID 10348466
- [Background] Little KY, Gorebig J, Carroll FI, Mapili J, Meador-Woodruff JH. Lack of dopamine receptor agonists effect on striatal dopamine transporter binding sites. Brain Res. 1996 Dec 2;742(1-2):313-6. doi: 10.1016/s0006-8993(96)01033-5. PMID 9117410
- [Background] Marek K, Innis R, van Dyck C, Fussell B, Early M, Eberly S, Oakes D, Seibyl J. [123I]beta-CIT SPECT imaging assessment of the rate of Parkinson's disease progression. Neurology. 2001 Dec 11;57(11):2089-94. doi: 10.1212/wnl.57.11.2089. PMID 11739831
- [Background] Morrish PK, Rakshi JS, Bailey DL, Sawle GV, Brooks DJ. Measuring the rate of progression and estimating the preclinical period of Parkinson's disease with [18F]dopa PET. J Neurol Neurosurg Psychiatry. 1998 Mar;64(3):314-9. doi: 10.1136/jnnp.64.3.314. PMID 9527140
- [Background] Nurmi E, Bergman J, Eskola O, Solin O, Hinkka SM, Sonninen P, Rinne JO. Reproducibility and effect of levodopa on dopamine transporter function measurements: a [18F]CFT PET study. J Cereb Blood Flow Metab. 2000 Nov;20(11):1604-9. doi: 10.1097/00004647-200011000-00010. PMID 11083235
- [Background] Parkinson Study Group. Dopamine transporter brain imaging to assess the effects of pramipexole vs levodopa on Parkinson disease progression. JAMA. 2002 Apr 3;287(13):1653-61. doi: 10.1001/jama.287.13.1653. PMID 11926889
- [Background] Fahn S; Parkinson Study Group. Does levodopa slow or hasten the rate of progression of Parkinson's disease? J Neurol. 2005 Oct;252 Suppl 4:IV37-IV42. doi: 10.1007/s00415-005-4008-5. PMID 16222436
- [Background] Rioux L, Frohna PA, Joyce JN, Schneider JS. The effects of chronic levodopa treatment on pre- and postsynaptic markers of dopaminergic function in striatum of parkinsonian monkeys. Mov Disord. 1997 Mar;12(2):148-58. doi: 10.1002/mds.870120204. PMID 9087972
- [Background] Schapira AH. Dopamine agonists and neuroprotection in Parkinson's disease. Eur J Neurol. 2002 Nov;9 Suppl 3:7-14. doi: 10.1046/j.1468-1331.9.s3.9.x. PMID 12464116
- [Background] Whone AL, Watts RL, Stoessl AJ, Davis M, Reske S, Nahmias C, Lang AE, Rascol O, Ribeiro MJ, Remy P, Poewe WH, Hauser RA, Brooks DJ; REAL-PET Study Group. Slower progression of Parkinson's disease with ropinirole versus levodopa: The REAL-PET study. Ann Neurol. 2003 Jul;54(1):93-101. doi: 10.1002/ana.10609. PMID 12838524
- [Background] Wooten GF. Agonists vs levodopa in PD: the thrilla of whitha. Neurology. 2003 Feb 11;60(3):360-2. doi: 10.1212/wnl.60.3.360. No abstract available. PMID 12578913